CLINICAL TRIAL: NCT00858845
Title: Clonidine and the Skeletal Myopathy of Heart Failure
Brief Title: Using Clonidine to Improve Leg Weakness in People With Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Holly R Middlekauff, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 641; R01HL084525 (NIH); NCT01046344 (obsolete NCT alias); NCT01826643 (obsolete NCT alias)
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Results first posted 2013-09-09 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure
Keywords: Leg Weakness; Skeletal Myopathy; Sympathetic Nerve Activity
MeSH Terms: conditions — Heart Failure | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clonidine patch (Experimental): Participants assigned to wear a clonidine patch.
  Interventions: Drug: Clonidine Patch
- Placebo (Placebo Comparator): Participants assigned to wear a matching placebo patch.
  Interventions: Other: Matching Placebo Patch

INTERVENTIONS:
Drug: Clonidine Patch — A clonidine patch (0.1 mg/week) to be worn for a period of 3 months.
  Other Names: Catapres-TTS
  Arms: Clonidine patch
Other: Matching Placebo Patch — A matching placebo patch to be worn for a period of 3 months.
  Arms: Placebo

SUMMARY:
People with heart failure often have weakness in their leg muscles. This study will determine whether the leg weakness is due to very high adrenaline levels and whether the medication clonidine can improve leg weakness.

DETAILED DESCRIPTION:
Heart failure is a common condition, affecting approximately 5 million people in the United States. People with heart failure are encouraged to exercise and lose weight. However, many people with heart failure develop weakness in their leg muscles, which can make exercise difficult. Increased sympathetic nerve activity, which involves the nerves that carry adrenaline, also occurs in people with heart failure. It is possible that the increased sympathetic nerve activity may actually cause the leg muscle weakness. Clonidine, a medication used to treat high blood pressure, has been found to decrease sympathetic nerve activity. This study will further examine the connection between leg weakness and sympathetic nerve activity. It will also evaluate the effectiveness of clonidine at decreasing leg weakness in people with heart failure. Results from this study may explain why some people with heart failure are unable to exercise and may help to identify ways in which leg strength can be increased.

This study will enroll people with heart failure. Participants will be randomly assigned to wear either a clonidine patch or a placebo patch for 3 months. Participants will wear the patch on their upper arm, and they will replace the patch each week. At study visits at baseline and Month 3, participants will undergo the following procedures:

* Sympathetic nerve activity recording, which will record nerve activity in the lower leg, using small electrodes inserted through the skin
* Muscle biopsy, in which a small piece of muscle tissue will be obtained from participants' legs
* Heart rate and blood pressure measurements
* Arterial baroreceptor measurements, in which the nerves in the body that respond to changes in blood pressure will be examined while participants receive different medications to increase and decrease their blood pressure
* Echocardiography to obtain images of the heart
* Magnetic resonance scan of the leg
* Passive exercise procedure, in which study researchers will conduct an arm exercise with participants

There will be no follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure

Exclusion Criteria:

* Currently on Coumadin therapy
* Experienced a heart attack in the 3 months before study entry
* Medically unable to receive clonidine
* Advanced kidney or liver disease

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly R. Middlekauff, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles Medical Center, Los Angeles, California, United States

REFERENCES:
- [Result] Middlekauff HR, Verity MA, Horwich TB, Fonarow GC, Hamilton MA, Shieh P. Intact skeletal muscle mitochondrial enzyme activity but diminished exercise capacity in advanced heart failure patients on optimal medical and device therapy. Clin Res Cardiol. 2013 Aug;102(8):547-54. doi: 10.1007/s00392-013-0564-3. Epub 2013 Apr 11. PMID 23575739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All heart failure patients were recruited from the Ahmanson-University of California, Los Angeles (UCLA) Cardiomyopathy Center between 2008-2011.
Pre-assignment Details: Of 44 heart failure patients interested, 25 were ineligible (medication changes (6), "too well" with either left ventricular ejection fraction(LVEF) >35% (3) or New York Heart Association (NYHA) Class I (2), transportation issues (4), morbidly obese (3), enrolled in exercise program (2), other (5)), and of the remaining 19 patients, 8 declined.
Groups:
- Clonidine Patch: Participants were assigned to wear a clonidine patch (0.1 mg/weekly) for a treatment period of 3 months.
- Placebo: Participants were assigned to wear a matching placebo patch (weekly) for a treatment period of 3 months.
Period: Overall Study
Arm/Group | Clonidine Patch | Placebo
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1
Not completed — Patient underwent heart transplant. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Patch: Participants were assigned to wear a matching placebo patch (0.1 mg/weekly) for a treatment period of 3 months.
- Total: Total of all reporting groups
Arm/Group | Clonidine Patch | Placebo Patch | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | NA — Data were not retained with detail needed to report by treatment arm. | NA — Data were not retained with detail needed to report by treatment arm | 4
  Male | NA — Data were not retained with detail needed to report by treatment arm | NA — Data were not retained with detail needed to report by treatment arm | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Citrate Synthase Activity as an Estimate of Mitochondrial Activity
Time Frame: Baseline, 3 months
Population: One patient randomized to placebo underwent urgent orthotopic heart transplantation before second measure could be obtained.
Measure: Mean (Standard Error); unit: micromole/min/wet weight
Arm/Group | Clonidine Patch | Placebo
Number analyzed (Participants) | 5 | 5
micromole/min/wet weight | -0.3 (0.09) | 0.07 (0.07)

2. Secondary Outcome: Change in Proportion of Type 1 Fibers
Description: Fibers were typed as I or II according to presence of myosin heavy chain.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of fibers
Arm/Group | Clonidine Patch | Placebo
Number analyzed (Participants) | 5 | 5
percentage of fibers | -4.6 (3.8) | -5.6 (1.9)

3. Other Pre Specified Outcome: Change in Muscle Sympathetic Nerve Activity
Description: Muscle sympathetic nerve activity was measured as bursts sympathetic nerve activity per minute.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: bursts/min
Arm/Group | Clonidine Patch | Placebo
Number analyzed (Participants) | 5 | 5
bursts/min | -4.3 (2.4) | 4.4 (8.8)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Clonidine Patch | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

LIMITATIONS AND CAVEATS:
This is a small trial, but it was not terminated early, and there were no technical issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes